CLINICAL TRIAL: NCT03182855
Title: Cangrelor vs. Ticagrelor for Early Platelet Inhibition in ST-elevation Myocardial Infarction
Brief Title: Cangrelor vs. Ticagrelor for Early Platelet Inhibition in STEMI
Acronym: CanTi
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Jacob Sørensen, Md, PhD, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-003721-41
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; STEMI - ST Elevation Myocardial Infarction
Keywords: Acute Coronary Syndrome; STEMI; Platelet reactivity; Anti-thrombotic therapy
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Ticagrelor; cangrelor

STUDY DESIGN:
Intervention Model Description: Randomized trial. No blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prehospital ticagrelor (Active Comparator): Ticagrelor 180 mg orally administered in the ambulance as soon as possible after inclusion and before coronary angiography. The two pills are chewed and swallowed with a glass of water.
  In both groups heparin and bivalirudin will be administered as part of routine therapy. In hemodynamically compromised patients with a high thrombus load a glycoprotein IIb/IIIa inhibitor may be used as bail-out therapy (these patients will be excluded). These drugs are not deemed to be study medication.
  Interventions: Drug: Ticagrelor
- Inhospital cangrelor tetrasodium (Active Comparator): Ticagrelor 180 mg orally in combination with cangrelor intravenously (bolus 30 μg/kg within 1 minute followed by infusion (4 μg/kg/minute) for two hours) both administered immediately after coronary angiography, when PPCI is indicated.
  In both groups heparin and bivalirudin will be administered as part of routine therapy. In hemodynamically compromised patients with a high thrombus load a glycoprotein IIb/IIIa inhibitor may be used as bail-out therapy (these patients will be excluded). These drugs are not deemed to be study medication.
  Interventions: Drug: Ticagrelor; Drug: Cangrelor Tetrasodium

INTERVENTIONS:
Drug: Ticagrelor — ADP-receptor blocker. Oral formulation. Standard Therapy in Acute Myocardial Infarction. Administered in the ambulance in arm 1 and in the hospital (catheterization laboratory) in arm 2.
  Other Names: Brilique; Brilinta
Drug: Cangrelor Tetrasodium — Intravenous ADP-receptor blocker. Administered after hospital arrival in the catheterization laboratory.
  Other Names: Kengrexal; Kengreal
  Arms: Inhospital cangrelor tetrasodium

SUMMARY:
This randomized, controlled trial compares the anti-thrombotic effect of cangrelor and ticagrelor on platelet activity in patients with acute ST-elevation myocardial infarction.

Patients will receive either prehospital ticagrelor (180 mg - crushed) or in-hospital cangrelor (bolus 30 μg/kg within 1 minute followed by infusion (4 μg/kg/minute) for two hours) followed by 180 mg ticagrelor.

The primary study end-point is platelet reactivity at sheath insertion, at the end of the PCI procedure (before sheath removal) and two hours after PCI is initiated. The secondary end-point is the proportion of patients with inappropriate or harmful P2Y12 administration.

DETAILED DESCRIPTION:
In patients with ST-elevation myocardial infarction (STEMI) early restoration of blood flow in the culprit coronary artery is essential to reduce infarct size and thereby mortality and morbidity. The recommended method for achieving reperfusion is primary percutaneous coronary intervention (PPCI) (1,2). Early initiation of adjunctive antithrombotic therapy is important to prevent further thrombus formation and to facilitate PPCI.

International guidelines currently recommend immediate oral or intravenous administration of aspirin and intravenous administration of heparin in patients with suspected STEMI (1,2).

A second platelet inhibitor (of the P2Y12 family) is often added already in the ambulance. This enhances the antiplatelet effect, but also increases bleeding risk.

A recently introduced antithrombotic agent, that can be administered intravenously, can potentially achieve the same antithrombotic effect at the same time of the oral agent, with the added benefit, that administration can await coronary angiography. This would reduce the risk of administrating powerful antithrombotic medicine to patients with diagnosis other than STEMI.

In the ATLANTIC trial (3) prehospital administration was compared to in-hospital (catheterization laboratory) administration of ticagrelor. The trial indicated that ticagrelor could safely be administered in the ambulance, although there was no apparent effect on Thrombolysis in Myocardial Infarction (TIMI) flow in the culprit coronary artery and no effect on ST-segment resolution in the ECG. However, the median time difference between ticagrelor administration in the two groups was only 31 minutes. This might not leave enough time for adequate platelet inhibition in the prehospital group.

In patients with NSTEMI (Non-ST-elevation myocardial infarction), pretreatment with prasugrel has been shown to be associated with increased bleeding risk and confers no benefit on ischemic outcomes (4). Thus, there are indications that the addition of oral P2Y12 inhibitor can await the coronary angiography, thereby minimizing the risk of excessive platelet inhibition in patients with a high bleeding risk or a potentially lethal differential diagnosis such as aortic dissection (5). Previous studies document that approximately 15% of patients with suspected STEMI have a final diagnosis other than an acute coronary syndrome (6). There is a fine balance between the benefit and possible deleterious effects of early, aggressive oral platelet inhibition in patients with suspected STEMI.

Recently a novel, intravenous P2Y12 inhibitor - cangrelor - has been released. Cangrelor enables immediate inhibition of the platelet P2Y12 inhibitor. The drug has a short half-life, is reversible and is only effective during administration (7). This contrasts with the available oral P2Y12 inhibitors, which all induce inhibition of the platelets for several days. Although ticagrelor is reversible, the platelet inhibition induced by this widely used, potent drug lasts for at least 3 days (8). The effects of cangrelor on platelet inhibition and clinical outcome have been documented in three, large clinical randomized trials (9-11).

Currently it is unknown whether platelet inhibition achieved by cangrelor administered in the catheterization laboratory is more effective compared to ticagrelor administered in the ambulance in patients with suspected STEMI.

The objective of this trial is to compare the effect of oral ticagrelor vs. intravenous cangrelor on platelet inhibition in ST-elevation myocardial infarction.

Patients will be included in the ambulance and randomized to one of two treatment groups; either to receive oral ticagrelor or intravenous cangrelor.

The study randomization will not be blinded to either investigator or patient (Open label, randomized, controlled clinical trial).

The hypothesis is that platelet inhibition with cangrelor administered intravenously in the catheterization laboratory after coronary angiography, but before PPCI is as effective as platelet inhibition achieved by ticagrelor administered orally in the ambulance in patients with suspected STEMI.

It is also assumed that administration of a P2Y12 inhibitor after coronary angiography reduces the proportion of inappropriate administration due to a final diagnosis other than STEMI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients triaged for PPCI due to suspicion of STEMI.
2. Symptom duration < 12 hours

Exclusion Criteria:

1. Previous inclusion in the study
2. Already in treatment with ticagrelor, prasugrel or clopidogrel
3. Treatment with oral anticoagulants (warfarin, coumarins, rivaroxaban, apixaban, dabigatran)
4. Adjunctive use of glycoprotein IIb/IIIa inhibitor during PCI
5. Active bleeding
6. Known, severe kidney failure (GFR < 30 ml/min) and/or liver disease
7. Women of child bearing ability who are not using contraceptive medication
8. Severe mental or psychiatric disease, altered mental state (including unconsciousness) making it impossible to achieve informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity 10 minutes PCI after is initiated | 10 minutes
  Platelet reactivity measured in platelet reactivity units (PRU) by the VerifyNow® assay 10 minutes after PCI is initiated.

SECONDARY OUTCOMES:
Platelet reactivity before and after PCI | 2 hours
  Effect on platelet reactivity, measured by VerifyNow® after sheath insertion, at the end of the PCI procedure (before sheath removal) and two hours after PCI is initiated
Proportion of patients with inappropriate or harmful P2Y12 administration | 4 hours
  This is defined as patients with a diagnosis other than acute myocardial infarction or patients where prehospital ticagrelor administration delays surgery (cardiac or other) due to excess bleeding risk.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob T Sorensen, MD, PhD, Principal Investigator — Aarhus University Hospital, Department of Cardiology, Skejby; Steen D Kristensen, MD, DMSc, Study Director — Aarhus University Hospital, Department of Cardiology, Skejby
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso JE, Tracy CM, Woo YJ, Zhao DX; CF/AHA Task Force. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2013 Jan 29;127(4):529-55. doi: 10.1161/CIR.0b013e3182742c84. Epub 2012 Dec 17. No abstract available. PMID 23247303
- [Background] Aradi D, Collet JP, Mair J, Plebani M, Merkely B, Jaffe AS, Mockel M, Giannitsis E, Thygesen K, ten Berg JM, Mueller C, Storey RF, Lindahl B, Huber K; Study Group on Biomarkers in Cardiology of the Acute Cardiovascular Care Association of the European Society of Cardiology; Working Group on Thrombosis of the European Society of Cardiology. Platelet function testing in acute cardiac care - is there a role for prediction or prevention of stent thrombosis and bleeding? Thromb Haemost. 2015 Feb;113(2):221-30. doi: 10.1160/TH14-05-0449. Epub 2014 Nov 20. PMID 25413597
- [Result] Montalescot G, van 't Hof AW, Lapostolle F, Silvain J, Lassen JF, Bolognese L, Cantor WJ, Cequier A, Chettibi M, Goodman SG, Hammett CJ, Huber K, Janzon M, Merkely B, Storey RF, Zeymer U, Stibbe O, Ecollan P, Heutz WM, Swahn E, Collet JP, Willems FF, Baradat C, Licour M, Tsatsaris A, Vicaut E, Hamm CW; ATLANTIC Investigators. Prehospital ticagrelor in ST-segment elevation myocardial infarction. N Engl J Med. 2014 Sep 11;371(11):1016-27. doi: 10.1056/NEJMoa1407024. Epub 2014 Sep 1. PMID 25175921
- [Result] Montalescot G, Bolognese L, Dudek D, Goldstein P, Hamm C, Tanguay JF, ten Berg JM, Miller DL, Costigan TM, Goedicke J, Silvain J, Angioli P, Legutko J, Niethammer M, Motovska Z, Jakubowski JA, Cayla G, Visconti LO, Vicaut E, Widimsky P; ACCOAST Investigators. Pretreatment with prasugrel in non-ST-segment elevation acute coronary syndromes. N Engl J Med. 2013 Sep 12;369(11):999-1010. doi: 10.1056/NEJMoa1308075. Epub 2013 Sep 1. PMID 23991622
- [Result] Hansson EC, Dellborg M, Lepore V, Jeppsson A. Prevalence, indications and appropriateness of antiplatelet therapy in patients operated for acute aortic dissection: associations with bleeding complications and mortality. Heart. 2013 Jan;99(2):116-21. doi: 10.1136/heartjnl-2012-302717. Epub 2012 Oct 9. PMID 23048167
- [Result] Becker S, Chisholm G, Maeng M. Positive predictive value of clinically suspected ST-segment elevation myocardial infarction using angiographic verification. Am J Cardiol. 2013 Oct 1;112(7):923-7. doi: 10.1016/j.amjcard.2013.05.026. Epub 2013 Jun 14. PMID 23768460
- [Result] Angiolillo DJ, Firstenberg MS, Price MJ, Tummala PE, Hutyra M, Welsby IJ, Voeltz MD, Chandna H, Ramaiah C, Brtko M, Cannon L, Dyke C, Liu T, Montalescot G, Manoukian SV, Prats J, Topol EJ; BRIDGE Investigators. Bridging antiplatelet therapy with cangrelor in patients undergoing cardiac surgery: a randomized controlled trial. JAMA. 2012 Jan 18;307(3):265-74. doi: 10.1001/jama.2011.2002. PMID 22253393
- [Result] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Result] Bhatt DL, Lincoff AM, Gibson CM, Stone GW, McNulty S, Montalescot G, Kleiman NS, Goodman SG, White HD, Mahaffey KW, Pollack CV Jr, Manoukian SV, Widimsky P, Chew DP, Cura F, Manukov I, Tousek F, Jafar MZ, Arneja J, Skerjanec S, Harrington RA; CHAMPION PLATFORM Investigators. Intravenous platelet blockade with cangrelor during PCI. N Engl J Med. 2009 Dec 10;361(24):2330-41. doi: 10.1056/NEJMoa0908629. PMID 19915222
- [Result] Harrington RA, Stone GW, McNulty S, White HD, Lincoff AM, Gibson CM, Pollack CV Jr, Montalescot G, Mahaffey KW, Kleiman NS, Goodman SG, Amine M, Angiolillo DJ, Becker RC, Chew DP, French WJ, Leisch F, Parikh KH, Skerjanec S, Bhatt DL. Platelet inhibition with cangrelor in patients undergoing PCI. N Engl J Med. 2009 Dec 10;361(24):2318-29. doi: 10.1056/NEJMoa0908628. PMID 19915221
- [Result] Bhatt DL, Stone GW, Mahaffey KW, Gibson CM, Steg PG, Hamm CW, Price MJ, Leonardi S, Gallup D, Bramucci E, Radke PW, Widimsky P, Tousek F, Tauth J, Spriggs D, McLaurin BT, Angiolillo DJ, Genereux P, Liu T, Prats J, Todd M, Skerjanec S, White HD, Harrington RA; CHAMPION PHOENIX Investigators. Effect of platelet inhibition with cangrelor during PCI on ischemic events. N Engl J Med. 2013 Apr 4;368(14):1303-13. doi: 10.1056/NEJMoa1300815. Epub 2013 Mar 10. PMID 23473369
- [Result] Parodi G, Xanthopoulou I, Bellandi B, Gkizas V, Valenti R, Karanikas S, Migliorini A, Angelidis C, Abbate R, Patsilinakos S, Baldereschi GJ, Marcucci R, Gensini GF, Antoniucci D, Alexopoulos D. Ticagrelor crushed tablets administration in STEMI patients: the MOJITO study. J Am Coll Cardiol. 2015 Feb 10;65(5):511-2. doi: 10.1016/j.jacc.2014.08.056. No abstract available. PMID 25660931
- [Result] Parodi G, Valenti R, Bellandi B, Migliorini A, Marcucci R, Comito V, Carrabba N, Santini A, Gensini GF, Abbate R, Antoniucci D. Comparison of prasugrel and ticagrelor loading doses in ST-segment elevation myocardial infarction patients: RAPID (Rapid Activity of Platelet Inhibitor Drugs) primary PCI study. J Am Coll Cardiol. 2013 Apr 16;61(15):1601-6. doi: 10.1016/j.jacc.2013.01.024. Epub 2013 Mar 22. PMID 23500251
- [Result] Alexopoulos D, Xanthopoulou I, Mavronasiou E, Stavrou K, Siapika A, Tsoni E, Davlouros P. Randomized assessment of ticagrelor versus prasugrel antiplatelet effects in patients with diabetes. Diabetes Care. 2013 Aug;36(8):2211-6. doi: 10.2337/dc12-2510. Epub 2013 Mar 14. PMID 23491524